CLINICAL TRIAL: NCT02216019
Title: Diagnostic Interest of Leukocyte Immunophenotyping Using Multiparameter 8-color Flow Cytometry in Heart Surgery
Acronym: INFLUX
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I13015 Influx
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; infectious complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study cohort: Patient undergoing planned heart surgery with cardiopulmonary bypass
  Interventions: Other: Whole blood

INTERVENTIONS:
Other: Whole blood — preoparatoire whole blood and postoperative whole blood

SUMMARY:
In septic patients, Septiflux1 study identified immature granulocytes which may have a diagnostic and prognostic interest. However, with these preliminary results it is not possible to make a difference between what is linked to the infection and what is a consequence of the inflammation which goes along with the septic process. Using flow cytometry, the study of leukocytes in a pure inflammatory model such as cardiopulmonary bypass in heart surgery could make possible to test the diagnostic interest of the immature granulocytes but also to attribute a prognostic value for the occurrence of post-operative infections.

DETAILED DESCRIPTION:
Expression of CD10, CD16, CD24, CD64 on granulocytes, of CD14 and CD16 on monocytes and of CD3 on T lymphocytes.

Flow cytometers will all be calibrated the same way using common reagents (known fluorescent calibration beads). Moreover, CD45 and CD3 level of expression on lymphocytes will help to check that the collection of data is standardized between the different centers.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient undergoing planned heart surgery with cardiopulmonary bypass

Exclusion Criteria:

* Pregnancy,
* progressive solid cancer,
* HIV infection,
* history of blood or inflammatory disease,
* long-term immunosuppressive treatment,
* urgent surgical intervention,
* documented preoperative infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing planned heart surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Expression of the marker CD64, CD10 and CD16 | 1 hour
  Evolution rate of CD64, CD10 and CD16 in the immediate postoperative cardiac surgery

SECONDARY OUTCOMES:
Early onset of infectious complications | 7 days
  Early onset of infectious complications in the 7 days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FRANCOIS, MD, Principal Investigator — CHU LIMOGES
Locations (1):
- CHU de Limoges - Service de réanimation polyvalente, Limoges, Limoges, France